CLINICAL TRIAL: NCT04783103
Title: Neuromodulation in the Elderly Depressed: a Brain Im-aging Pilot Study
Brief Title: Neuromodulation in the Elderly Depressed: a Brain Imaging Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Dieter Zeeuws, Dieter Zeeuws, MD, Head of Clinic in psychiatry, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020/324
Record Dates: First submitted 2021-02-15; First posted 2021-03-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Old Age; Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: In a sham-controlled randomized controlled trial, we will treat 44 geriatric depressed patients with accelerated dTMS (adTMS) (5 sessions/day over 4 days) and evaluate clinical efficacy and safety. One week after the last adTMS or sham treatment, all patients will have access to active treatment in a 3 week open label transcutaneous direct current stimulation (tDCS) with a home-use device. In this manner we can examine clinical effect of tDCS in the adTMS-sham group as well as the possible maintenance effect of tDCS in the adTMS active treatment group. Because newly introduced neuromodulation paradigms should go through profound neurobiological testing before applying them on a regular basis, this research will include multimodal brain imaging techniques to elucidate the working mechanisms of these applications in order to optimize response prediction and treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects will be assigned to one of the treatment arms by use of the top card from a stack of pre-coded cards which were prepared by an independent coder. The card has to be entered in machine in order to operate it and can be an activator of either sham or active treatment (both are integrated in and delivered by the same helmet coil.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active adTMS (Active Comparator): Subjects in the treatment arm receive 20 sessions of real adTMS . The sessions will be spread over the four succeeding days (5 sessions daily on Tuesday, Wednesday, Thursday and Friday).
  Interventions: Device: a Magstim Rapid2 Plus1 Magnetic Stimulator connected to a Brainsway H1 coil
- Sham adTMS (Sham Comparator): Subject in the control/Placebo/Sham arm receive 20 sessions of sham adTMS. The sessions will be spread over the four succeeding days (5 sessions daily on Tuesday, Wednesday, Thursday and Friday).
  Interventions: Device: a Magstim Rapid2 Plus1 Magnetic Stimulator connected to a Brainsway H1 coil

INTERVENTIONS:
Device: a Magstim Rapid2 Plus1 Magnetic Stimulator connected to a Brainsway H1 coil — 3 weeks home use
  Other Names: Sooma tDCS (open label)

SUMMARY:
To evaluate safety and efficacy of an accelerated deep brain Transcranial Magnetic stimulation (adTMS) and transcutaneous direct current stimulation (tDCS) protocol in an elderly depressed patient population

DETAILED DESCRIPTION:
With a growing number of elderly persons, geriatric depression - associated with important morbidity and mortality- is becoming a significant health problem. Given the risk of polypharmacy and increased side effects, alternative non pharmaceutical treatments such as repetitive transcranial magnetic stimulation (rTMS) and transcutaneous direct current stimulation (tDCS) may offer a solution. Given our recent positive results with accelerated rTMS in the elderly depressed, we want to continue to develop non-invasive treatment stimulations. The FDA approved deep brain TMS (dTMS) technique may be a promising option, targeting the brain underneath the neocortex with potentially better response and remission rates. Therefore, in a sham-controlled randomized controled trial, we will treat 44 geriatric depressed patients with accelerated dTMS (5 sessions/day over 4 days only), and evaluate clinical efficacy and safety. One week after the last adTMS or sham treatment, all patients will have access to active treatment in a 3 week open label transcutaneous direct current stimulation (tDCS) with a home-use device. In this manner we can examine clinnical effect of tDCS in the adTMS-sham group as well as the possible maintenance effect of tDCS in the adTMS active treatment group. Because new introduced neuromodulation paradigms should be rigorously neurobiologically examined before applying them on a regular basis, this research will include multimodal brain imaging techniques to elucidate the working mechanisms of these applications in order to optimize response prediction and treatment. Gut microbes can influence human metabolism, nutrition, physiology and immune status. The "microbiota-gut-brain axis" entails a continues exchange of information between the gut and central nervous system. Several clinical and preclinical studies have emphasized the bidirectional role of microbiome disruption in depression and depression-like behavior. In the current project, we also will examine the effects of neurostimulation treatments on the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* • In- and outpatients (age 65 year or older).

  * Meeting the Diagnostic and Statistical Manual of Mental Disorders (DSM 5) criteria for unipolar depression according 17-item Hamilton depression rating scale (HDRS-17) score of 17 or more.
  * Failed to respond to at least one adequate course with an antidepressant medication trial, including the current one.
  * Intention to continue the current (>6 weeks) antidepressant treatment at a stable dose dur-ing the stimulation.
  * Benzodiazepines are permitted up to a maximum dose of 40 mg diazepam or equivalent. If the dosage has been recently changed, it should be stable for at least 2 weeks.
  * Able to read, understand and sign the Informed Consent Form.

Exclusion Criteria:

* • Psychosis (except depression with psychotic features).

  * A personal history of seizures or epilepsy, a history of seizures or epilepsy in first degree relatives and the presence of any known factor that can lower the seizure threshold (sleep deprivation, substance abuse, etc.), previous head injury and the presence of metallic implants in the cephalic region (e.g., aneurysm clips, shunts, stimulators, cochlear implants, electrodes) with the exception of dental fillings. The presence of cardiac pacemakers, neurostimulators, surgical clips or other electronic equipment, comorbidity with the following neurological disorders: increased intracranial pressure, space-occupying lesion, history of stroke or transient ischemic attack, brain aneurysm and any structural brain damage with increased risk for epilepsy detected with (study related) MRI.
  * Patients with cognitive disturbances or dementia (Mini Mental State) < 24.
  * Suicide attempt within 6 months before the start of the study or present high risk of suicide per the investigator's clinical judgment and indicative response* on the Columbia-Suicide Severity Rating Scale (C-SSRS) and 21-items Beck Scale for Suicide Ideation (BSI). *'yes' on Item 5 (active suicidal ideation with specific plan and intent).
  * Any change in the habitual psychopharmacological agents will be considered as dropout.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical effect of adTMS (Changes in depression severity clinician-rated and self-report) | screening, Day 1 (+/-3d), Day 8 (+/-3d) ,Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the effect of adTMS delivered by a H1 coil to the left Dorsolateral Prefrontal Cortex (DLPFC), as an add-on treatment, on depressive symptoms in a sample of elderly patients with MDD.-measured by change in the 17 item Hamilton Depression rating Scale score. For a total score between 0 and 48, the higher the total score the more severe the depression. Response is reduction from baseline of ≥ 50% in the total score and remission is a total HAMD-17 score ≤ 7.
  * measured by change in the Beck-Inventory of Depression-II score. For a total score between 0 and 63, the higher the total score the more severe the depression. A score of ≤9 is the criterion for remission and BDI-II score decrease of 50% from baseline is the criterion for treatment response.
  * measured by change in the Geriatric Depression Scale 15 item version (GDS-15) self-rating scale score.

SECONDARY OUTCOMES:
Clinical effect of tDCS 17 item Hamilton Depression rating Scale score | Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the effect of tdCS delivered by a Sooma tDCS to the left Dorsolateral Prefrontal Cortex (DLPFC), as an add-on treatment, on depressive symptoms in a sample of elderly patients with MDD.-measured by change in the 17 item Hamilton Depression rating Scale score. For a total score between 0 and 48, the higher the total score the more severe the depression. Response is reduction from baseline of ≥ 50% in the total score and remission is a total HAMD-17 score ≤ 7.
Clinical effect of tDCS Beck-Inventory of Depression-II score | Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the effect of tdCS delivered by a Sooma tDCS to the left Dorsolateral Prefrontal Cortex (DLPFC), as an add-on treatment, on depressive symptoms in a sample of elderly patients with MDD.-measured by change in the Beck-Inventory of Depression-II score. For a total score between 0 and 63, the higher the total score the more severe the depression. A score of ≤9 is the criterion for remission and BDI-II score decrease of 50% from baseline is the criterion for treatment response.
Clinical effect of tDCS Geriatric Depression Scale 15 item version (GDS-15) self-rating scale score | Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the effect of tdCS delivered by a Sooma tDCS to the left Dorsolateral Prefrontal Cortex (DLPFC), as an add-on treatment, on depressive symptoms in a sample of elderly patients with MDD.-measured by change in the Geriatric Depression Scale 15 item version (GDS-15) self-rating scale score. Score of ≤6 is the criterion for remission and decrease of 50% from baseline is the criterion for treatment response.
maintenance effect of tDCS 17 item Hamilton Depression rating Scale score | Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the maintenance effect of tdCS delivered by a Sooma tDCS to the left Dorsolateral Prefrontal Cortex (DLPFC), as an add-on treatment, on depressive symptoms in a sample of elderly patients with MDD who responded to active adTMS measured by reduction from baseline of ≥ 50% in the total score in the 17 item Hamilton Depression rating Scale score. Maintenance effect occurs if the responders scores at day 15 remain or are lower on day 36.
maintenance effect of tDCS Beck-Inventory of Depression-II score | Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the maintenance effect of tdCS delivered by a Sooma tDCS to the left Dorsolateral Prefrontal Cortex (DLPFC), as an add-on treatment, on depressive symptoms in a sample of elderly patients with MDD who responded to active adTMS measured by reduction from baseline of ≥ 50% in the total score in the BDI-II score decrease of 50% from baseline in the Beck-Inventory of Depression-II score. Maintenance effect occurs if the responders scores at day 15 remain or are lower on day 36.
functional magnetic resonance imaging changes pre/post treatment in gender task as an incidental measure of emotional processing and probe of limbic function, and it's predictive value for response | Day 1 (+/-3d), Day 8 (+/-3d)
  To investigate if the fMRI gender task provides an incidental measure of emotional processing and could be a better probe of limbic function, and it's predictive value for response to adTMS and/or tDCS.To look for change post-pre intervention in the fMRI gender task response.
effect on cognition MMSE | screening, Day 8 (+/-3d) ,Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the effect of adTMS and tDCS on cognition as measured by increase in Mini Mental State examination scores.Scores range from 0 to 30, a score increase indicates improvement.
Incidence of Treatment-Emergent Adverse Events assessed with the Adverse Events questionnaire | Day 8 (+/-3d) ,Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the safety profile of adTMS and tDCS for elderly with MDD
effect on suicide risk as measured by change in C-SSRS | screening, Day 1 (+/-3d), Day 8 (+/-3d) ,Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the effect of adTMS and tDCS on suicide risk of elderly patients with MDD.
effect on suicide risk as measured by change in BSI | screening, Day 1 (+/-3d), Day 8 (+/-3d) ,Day 15 (+/-3d) Day 36 (+/-3d)
  To investigate the effect of adTMS and tDCS on suicide risk of elderly patients with MDD.
effect on the gut microbiome | Day 1 (+/-3d), Day 8 (+/-3d) Day 36 (+/-3d)
  To investigate the effect of neurostimulation on the gut microbiome in elderly with MDD.
possible neuroimaging biological markers for response | Day 1 (+/-3d), Day 8 (+/-3d) Day 36 (+/-3d)
  To investigate possible neurobiological markers for response to adTMS and/or tDCS by neuro imaging changes after adTMS and/or tDCS compared to baseline. Pre/Post changes in resting state fMRI en ASL (bloodflow) images.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Zeeuws, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All data will be disclosed after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of results
Access Criteria: research